CLINICAL TRIAL: NCT01632683
Title: Comparative Effectiveness of the C-MAC D-blade to Glidescope Videolaryngoscope in the Predicted Difficult Airway
Brief Title: STorz Against Glidescope Effectiveness
Acronym: STAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Iowa (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Michael Aziz, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 62199040
Record Dates: First submitted 2012-06-14; First posted 2012-07-03 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-10

CONDITIONS: Difficult Airway
Keywords: difficult airway; video laryngoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C-MAC (Active Comparator): Providers will utilize the C-MAC video laryngoscope equipped with a D-blade to facilitate intubation
  Interventions: Device: C-MAC
- Glidescope (Active Comparator): Providers will utilize the Glidescope video laryngoscope equipped with the #4 blade to facilitate intubation
  Interventions: Device: Glidescope

INTERVENTIONS:
Device: C-MAC — C-MAC arm
  Arms: C-MAC
Device: Glidescope — Glidescope arm
  Arms: Glidescope

SUMMARY:
This study evaluates success rates of tracheal intubation (passing a breathing tube)for patients who may be more challenging to intubate while utilizing one of two devices that facilitate placement of the tube with video technology.

ELIGIBILITY:
Inclusion Criteria:

* adult 18 years of age
* Mallampati classification scale score of 3 or 4
* Neck circumference greater than 40cm for males, 38 cm for females
* mouth opening less than 3cm, but greater than 2cm

Exclusion Criteria:

* children
* prisoners
* history of easy intubation (success on first attempt with direct laryngoscopy)
* known unstable cervical spine injury
* emergency surgery
* nasal intubation route
* planned awake technique

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Aziz MF, Dillman D, Fu R, Brambrink AM. Comparative effectiveness of the C-MAC video laryngoscope versus direct laryngoscopy in the setting of the predicted difficult airway. Anesthesiology. 2012 Mar;116(3):629-36. doi: 10.1097/ALN.0b013e318246ea34. PMID 22261795

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | C-MAC | Glidescope
Started | 548 | 552
Completed | 548 | 552
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | C-MAC | Glidescope | Total
Number analyzed (Participants) | 548 | 552 | 1100
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (13.7) | 54.4 (14.1) | 53.7 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 292 | 267 | 559
  Male | 256 | 285 | 541

OUTCOME MEASURES:

1. Primary Outcome: Intubation Success Rate
Description: Success rate is defined as a single blade insertion with successful tracheal tube placement confirmed by return of end-tidal carbon dioxide
Time Frame: 1 week
Measure: Number; unit: participants
Arm/Group | C-MAC | Glidescope
Number analyzed (Participants) | 548 | 552
participants | 512 | 531

2. Secondary Outcome: Intubation Time
Description: Intubation time is defined as the time from blade insertion to first return of end-tidal carbon dioxide
Time Frame: 1 week
Measure: Mean (Inter-Quartile Range); unit: seconds
Arm/Group | C-MAC | Glidescope
Number analyzed (Participants) | 548 | 552
seconds | 47 [39 to 60] | 47 [38 to 58]

3. Secondary Outcome: Graded Score of Laryngeal View Achieved
Description: Laryngeal view is defined by the modified Cormack and Lehane scale (1-4) and is assessed by the clinician and the study team. Grade 1 is considered to be a good view while grade 4 is considered to be a poor view.
Time Frame: 1 week
Population: Cormack-Lehane grade
Measure: Number; unit: participants
Units Other Than Participants: grade
Arm/Group | C-MAC | Glidescope
Number analyzed (Participants) | 541 | 557
Number analyzed (grade) | 4 | 4
participants
  Grade 1 | 482 | 398
  Grade 2 | 41 | 146
  Grade 3 | 8 | 11
  Grade 4 | 10 | 2

4. Secondary Outcome: Number of Particpants Requiring Adjuncts to Assist Intubation
Description: The need for use of a gum-elastic bougie or external laryngeal manipulation to facilitate tube placement will be measured by the study team.
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | C-MAC | Glidescope
Number analyzed (Participants) | 548 | 552
Participants | 117 | 128

5. Secondary Outcome: Number of Participants With Observed Complications
Description: Patients will be examined for evidence of mucosal or dental injury upon intervention. Patients will be asked if they have a sore throat in the recovery room, and their medical record will be reviewed to determine if any other airway related complications were observed by the clinical team including the need for reintubation or steroid administration to reduce swelling.
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | C-MAC | Glidescope
Number analyzed (Participants) | 548 | 552
Participants | 97 | 85

ADVERSE EVENTS:
Arm/Group | C-MAC | Glidescope
Serious Adverse Events (participants affected / at risk) | 0/548 | 0/552
Other Adverse Events (participants affected / at risk) | 4/548 | 7/552
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C-MAC (N=548) | Glidescope (N=552)
pharyngeal injury (Surgical and medical procedures) | 4 | 7 — pharyngeal injury

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No